CLINICAL TRIAL: NCT02967237
Title: An Interventional, Open-label, Single-arm, Multicenter, 24 Weeks Phase 4 Study Assessing the Efficacy and Safety of Toujeo in Patients With Type 2 Diabetes Inadequately Controlled With Basal Insulin
Brief Title: Evaluation of Toujeo Insulin in Type 2 Diabetes Patients Inadequately Control With Their Basal Insulin Treatment
Acronym: Transition II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLARGL07667; 2015-002416-33 (EudraCT Number); U1111-1176-6203 (Other: UTN)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin glargine (U300) (Experimental): Type 2 diabetes mellitus patients uncontrolled with their current basal insulin therapy switched according to the physician decision, to insulin glargine (U300) administered subcutaneously and once daily using a pre-filled pen
  Interventions: Drug: insulin glargine (U300)

INTERVENTIONS:
Drug: insulin glargine (U300) — Pharmaceutical form: solution Route of administration: subcutaneous
  Other Names: HOE901; Toujeo

SUMMARY:
Primary Objective:

The primary objective is to describe the effect of insulin glargine (U300) in type 2 diabetes mellitus (T2DM) patients uncontrolled with their current basal insulin therapy and eligible for basal switching, according to the Physician decision, on glycated hemoglobin (HbA1c) improvement.

Secondary Objectives:

* Evolution of fasting plasma glucose
* Evolution of insulin dose and body weight
* Hypoglycemia incidence
* Safety
* Patients satisfaction when they change their insulin for HOE901-U300

DETAILED DESCRIPTION:
The total study duration per patient is approximately 28 weeks.

ELIGIBILITY:
Inclusion criteria :

* Type 2 diabetic adult patients treated with basal insulin, with or without oral anti-diabetic agents, with or without glucagon-like peptide-1 (GLP-1) receptor agonist
* HbA1c > 7.5%

Exclusion criteria:

* Patients with high dose of insulin (>1.2 U/kg)
* Use of prandial insulin
* Change of dose of antidiabetic drugs within the last 8 weeks
* Use of systemic glucocorticoids during at least 2 weeks in the last 12 weeks

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-01-04; Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1c | Baseline, Week 24

SECONDARY OUTCOMES:
Percentage of patients who reach target fasting plasma glucose (90-130 mg/dL) | At Weeks 12 and 24
Percentage of patients with HbA1c <7%, <7.5%, and <8% | At Week 24
Mean change from baseline in HbA1c across HbA1c subgroups category (≤8%, >8 to 9%, and >9%) | Baseline to Week 12 and Week 24
Mean change from baseline in fasting plasma glucose | Baseline to Week 12 and Week 24
Assessment of patient reported outcomes (satisfaction on treatment and perception of hypoglycemia/hyperglycemia) based on the Diabetes Treatment Satisfaction Questionnaire (DTSQ) | Baseline to Week 24
Change in Diabetes Treatment Satisfaction Questionnaire score | Week 24
Number of hypoglycemic events | From inclusion up to Week 24
Number of adverse events | From inclusion up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (85):
- France (85):
  - Investigational Site Number 250017, Alençon
  - Investigational Site Number 250073, Alès
  - Investigational Site Number 250047, Amiens
  - Investigational Site Number 250028, Amilly
  - Investigational Site Number 250062, Bagnols-sur-Cèze
  - Investigational Site Number 250093, Bar-le-Duc
  - Investigational Site Number 250020, Besançon
  - Investigational Site Number 250081, Béthune
  - Investigational Site Number 250034, Bondy
  - Investigational Site Number 250022, Brest
  - Investigational Site Number 250070, Brest
  - Investigational Site Number 250060, Cahors
  - Investigational Site Number 250096, Cannes
  - Investigational Site Number 250072, Chambéry
  - Investigational Site Number 250037, Châlons-en-Champagne
  - Investigational Site Number 250018, Cholet
  - Investigational Site Number 250068, Clermont-Ferrand
  - Investigational Site Number 250098, Cognac
  - Investigational Site Number 250048, Colmar
  - Investigational Site Number 250088, Contamines Sur Arve
  - Investigational Site Number 250054, Coudray
  - Investigational Site Number 250063, Dijon
  - Investigational Site Number 250013, Eaubonne
  - Investigational Site Number 250095, Étampes
  - Investigational Site Number 250104, Grenoble
  - Investigational Site Number 250004, La Roche-sur-Yon
  - Investigational Site Number 250002, La Rochelle
  - Investigational Site Number 250019, La Seyne-sur-Mer
  - Investigational Site Number 250030, Lamagistère
  - Investigational Site Number 250103, Le Chesnay
  - Investigational Site Number 250053, Le Creusot
  - Investigational Site Number 250044, Le Mans
  - Investigational Site Number 250056, Lens
  - Investigational Site Number 250051, Lourdes
  - Investigational Site Number 250071, Mantes-la-Jolie
  - Investigational Site Number 250092, Marseille
  - Investigational Site Number 250064, Marseille
  - Investigational Site Number 250089, Maubeuge
  - Investigational Site Number 250083, Mérignac
  - Investigational Site Number 250035, Montpellier
  - Investigational Site Number 250061, Montpellier
  - Investigational Site Number 250010, Montpellier
  - Investigational Site Number 250008, Montpellier
  - Investigational Site Number 250032, Mulhouse
  - Investigational Site Number 250043, Nancy
  - Investigational Site Number 250005, Narbonne
  - Investigational Site Number 250069, Nevers
  - Investigational Site Number 250052, Nîmes
  - Investigational Site Number 250059, Noisy-le-Grand
  - Investigational Site Number 250058, Orléans
  - Investigational Site Number 250031, Paris
  - Investigational Site Number 250105, Paris
  - Investigational Site Number 250086, Paris
  - Investigational Site Number 250026, Paris
  - Investigational Site Number 250101, Pessac
  - Investigational Site Number 250084, Périgueux
  - Investigational Site Number 250107, Pointe à Pitre
  - Investigational Site Number 250067, Pontoise
  - Investigational Site Number 250078, Pringy
  - Investigational Site Number 250042, Reims
  - Investigational Site Number 250012, Roubaix
  - Investigational Site Number 250055, Roubaix
  - Investigational Site Number 250102, Saint-Brieuc
  - Investigational Site Number 250065, Saint-Denis
  - Investigational Site Number 250029, Saint-Mandé
  - Investigational Site Number 250108, Saint-Pierre
  - Investigational Site Number 250087, Seclin
  - Investigational Site Number 250090, Sète
  - Investigational Site Number 250006, Strasbourg
  - Investigational Site Number 250024, Strasbourg
  - Investigational Site Number 250033, Suresnes
  - Investigational Site Number 250057, Tarbes
  - Investigational Site Number 250001, Toulouse
  - Investigational Site Number 250076, Toulouse
  - Investigational Site Number 250082, Toulouse
  - Investigational Site Number 250050, Toulouse
  - Investigational Site Number 250027, Tours
  - Investigational Site Number 250075, Tours
  - Investigational Site Number 250041, Valenciennes
  - Investigational Site Number 250021, Vandœuvre-lès-Nancy
  - Investigational Site Number 250023, Vénissieux
  - Investigational Site Number 250039, Vichy
  - Investigational Site Number 250046, Vichy
  - Investigational Site Number 250100, Villeneuve-sur-Lot
  - Investigational Site Number 250007, Warloy-Baillon

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org